CLINICAL TRIAL: NCT04838002
Title: Comparative Effects of Radial and Focused Extracorporeal Shock Wave Therapies on Lateral Epicondylitis: A Randomised Sham-controlled Trial
Brief Title: The Effects of Radial and Focused Extracorporeal Shock Wave Therapies on Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şeyhmus KAPLAN (Other)
Responsible Party: Sponsor-Investigator, Şeyhmus KAPLAN, Principal Investigator, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yuzuncu Yil University Turkey
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Lateral Epicondylitis; Pain
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focus ESWT (Active Comparator)
  Interventions: Device: Extracorporeal shock wave
- Radial ESWT (Active Comparator)
  Interventions: Device: Extracorporeal shock wave
- Sham ESWT (Sham Comparator)
  Interventions: Device: Extracorporeal shock wave

INTERVENTIONS:
Device: Extracorporeal shock wave — Focus and Radial types Extracorporeal shock wave therapy

SUMMARY:
To date, focused and radial types of extracorporeal shock wave therapy have been effectively used in lateral epicondylitis. However, studies directly addressing a comparison between radial and focused types of extracorporeal shock wave therapy in lateral epicondylitis have not been done. Therefore, this study aims to evaluate comparative effects of radial and focused extracorporeal shock wave therapy options on lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lateral epicondylitis
* be aged ≥18 at the time of diagnosis
* be give informed consent

Exclusion Criteria:

* be have not completed the assessment process.
* elbow deformity
* psychological illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 min.
  pain evaluation, higher scores mean a worse outcome.
Patient-Rated Tennis Elbow Evaluation | 5 min.
  Scale, Higher scores represent higher level of pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyhmus Kaplan, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No